CLINICAL TRIAL: NCT04077905
Title: A Prospective Study on the Modified DEP Regimen Induction Therapy in Lymphoma Induced Hemophagocytic Lymphohistiocytosis
Brief Title: Pegylated Liposomal Doxorubicin as a Induction Therapy for Lymphoma Induced Hemophagocytic Lymphohistiocytosis.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Principal Investigator, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DMS-HLH-01
Record Dates: First submitted 2019-08-31; First posted 2019-09-04 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Hemophagocytic Lymphohistiocytosis
Keywords: pegylated liposomal doxorubicin
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — liposomal doxorubicin; Etoposide; Methylprednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DEP regimen (Experimental): pegylated liposomal doxorubicin, etoposide and methylprednisolone administered in 2 week cycles for 2 cycles
  Interventions: Drug: Pegylated liposomal doxorubicin; Drug: Etoposide; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Pegylated liposomal doxorubicin — 35mg/m² ivgtt on day 1
Drug: Etoposide — 100mg/m² ivgtt on day 1
Drug: Methylprednisolone — 2 mg/kg ivgtt or PO days 1 to 3, 0.75 mg/kg ivgtt or PO days 4 to 7, 0.25 mg/kg ivgtt or PO days 8 to 10, 0. 1 mg/kg ivgtt or PO days 11 to 14,

SUMMARY:
This study aimed to investigate the efficacy and safety of pegylated liposomal doxorubicin together with etoposide and methylprednisolone as a induction therapy for lymphoma induced hemophagocytic lymphohistiocytosis.

ELIGIBILITY:
Inclusion Criteria:

* 1.Diagnosed as lymphoma-Hemophagocytic Lymphohistiocytosis.
* 2.Patients were older than 2 years of age.
* 3.Estimated survival time ≥ 1 week.
* 4.Cardiac ultrasound LVEF≥50%; No Active bleeding of the internal organs(digestive tract, lung, brain, etc.); If the patient has dyspnea, oxygenation index >250.
* 5.sign informed consent.

Exclusion Criteria:

* 1.Heart function above grade II (NYHA).
* 2.Accumulated dose of doxorubicin above 400mg/m2 、epirubicin above 750mg/m2、pirarubicin above 800mg/m2 or the patients treated with anthracycline induced cardiovascular disease.
* 3.Pregnancy or lactating Women.
* 4.Allergic to pegylated liposomal doxorubicin or etoposide.
* 5.Active bleeding of the internal organs.
* 6.HIV antibody positivity.
* 7.Acute or chronic active hepatitis B (HBsAg positivity, HBV DNA negative acceptable), acute or chronic active hepatitis C (HCV antibody negatively acceptable; HCV antibody positivity, HCV RNA negative acceptable).
* 8.Participate in other clinical research at the same time.
* 9.The researchers considered that patients are not suitable for the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-08-31 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Response rate | Time Frame: 1 years
  complete response (CR) and partial response (PR) rates

SECONDARY OUTCOMES:
Response rate of lymphoma | Time Frame: 1 years
  complete response (CR) and partial response (PR) rates, using the standard response criteria (Cheson and al.)
Progression Free Survival | Time Frame: 1 years
  from date of inclusion to date of progression, relapse, or death from any cause Overall Survival
Overall Survival | Time Frame: 1 years
  from the date of inclusion to date of death, irrespective of cause Adverse Events
Adverse Events | Time Frame: 1 years
  any unfavorable and unintended sign , symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pi Y, Wang J, Zhou H, Ye X, Sun X, Liu L, Pan X, Wang Z. Modified DEP regimen as induction therapy for lymphoma-associated hemophagocytic lymphohistiocytosis: a prospective, multicenter study. J Cancer Res Clin Oncol. 2023 Jul;149(7):3033-3041. doi: 10.1007/s00432-022-04157-0. Epub 2022 Jul 19. PMID 35852619